CLINICAL TRIAL: NCT04454931
Title: Evaluation of the Effect of Endotracheal Suctioning Applied at Different Head Height on Oxygenation of the Brain by Non-Invasive Method in Intensive Care Patients
Brief Title: Evaluation of the Effect of Endotracheal Suctioning Applied at Different Head Heights on the Oxygenation of the Brain
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Sibel Köstekli, Research Assistant, Zonguldak Bulent Ecevit University
Other Study IDs: 2019-19093093-01
Record Dates: First submitted 2020-03-04; First posted 2020-07-02 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Nurse's Role; Endotracheal Aspiration
Keywords: neurosurgery patient; endotracheal suctioning; nursing care; cerebral oxygenation; optimal head height

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Intensive care patients who underwent neurosurgery: Cerebral oxygenation status will be monitored during and after endotracheal suctioning in each patient included in the study. Non-invasive regional oximetry probes are placed in the frontal region of the patient and the patient will be positioned at the head height of 15 degrees with a 3-motor angle determining bearing system. Then, when the patient's need for endotracheal suctioning arises, endotracheal suctioning will be performed and the cerebral oxygenation status before the procedure, 1 minute, 5 minutes and 30 minutes after the procedure will be recorded on the monitor of the non-invasive regional oximeter device operating with NIRS technology. The same procedure will be applied to the patient at head heights of 30 and 45 degrees. Cerebral oxygenation status measured at each head height will be compared with appropriate statistical methods and the most appropriate head height will be determined.
  Interventions: Device: Root® with O3® Regional Oximetry

INTERVENTIONS:
Device: Root® with O3® Regional Oximetry — May help clinicians monitor cerebral oxygenation in situations in which pulse oximetry alone may not be fully indicative of the oxygen in the brain.
  It was aimed to determine the appropriate head height that should be given to patients in order to correct the endotracheal suctioning sequence, which is the most important care application of the neurosurgery patients who are followed up in the intensive care unit after surgery, and the possibility of subsequent disruption of cerebral perfusion. Therefore, cerebral oxygenation status, which is the most important parameter that shows the cerebral perfusion status of patients during and after the application, will be followed up by nurses with a non-invasive cerebral oximeter device.

SUMMARY:
In order for the brain, which is the most metabolically active organ of our body, to maintain its functions, it must reach oxygen saturation in the best way with continuous and rich blood flow.

Neurosurgery patients are followed for a while in the intensive care unit with a mechanical ventilator. During the care of the patient in mechanical ventilation; position changes, head height, endotracheal aspiration, oral care and invasive procedures that cause painful stimuli to the patient are factors that can affect brain perfusion pressure and oxygenation status of brain cells. It is known that high intracranial pressure, especially during and after endotracheal aspiration application, causes serious conditions in patients by disrupting cerebral blood flow.

It is also seen that cerebral blood flow is associated with head and body positions given in the postoperative period. It is stated in the literature that neurosurgical patients should be 30-45 degrees for proper head height in bed. In these patients, the height of the head should be in a suitable position for the correction of cerebral blood flow, which deteriorates during endotracheal aspiration, since autoregulation mechanisms are impaired or always activated. However, when the literature is examined, no information about the ideal head height that should be given to patients during endotracheal aspiration was found.

In addition, one of the most important parameters indicating the presence of cerebral complications is monitoring of cerebral oxygenation. It is stated that the most appropriate follow-up for patients should be evaluated by nurses in a non-invasive method.

In this study; In neurosurgery intensive care patients, endotracheal aspiration will be applied during endotracheal aspiration at head heights of 15, 30 and 45 degrees and it is aimed to determine the most appropriate head height during and after application by monitoring non-invasive cerebral oximeter device.

DETAILED DESCRIPTION:
Although the brain is only 2% of body weight,it is the most metabolically active and vital organ of the body.Cells in the brain; they need higher amounts of oxygen and energy than other organs in the body. Therefore, in order to maintain brain functions,rich and continuous blood flow and optimal oxygen saturation are required. Cerebral blood flow(SKA) is the most important factor in nutrition that provides oxygen saturation. Cerebral blood flow;Cerebral perfusion pressure(SPB) is affected by mean arterial pressure(MAP) and intracranial pressure(KIB).Under normal conditions, while SPB is constant, the conditions affecting blood pressure and cerebral venous return and elevation of KIB affect SPB.While normal cerebral blood flow is 50-70 ml/100 g/tissue/min;In cases where blood flow is interrupted,serious flow disruptions occur in cerebral circulation when the flow rate drops below 20 ml and vital conditions such as cerebral ischemia occur.

In cerebral blood flow intensive care patients;it may be disrupted during some maintenance procedures that cause painful stimuli such as position change,head height,endotracheal suctioning,oral care, and invasive procedures.In the literature;It is reported that if the cerebral blood flow drops below 20 ml/100 g/min for 30 minutes,it will reversibly stop the function of neurons,and if it falls below 10 ml/100 g/min for 30 minutes, irreversible neuron damage will occur.Therefore, in order to prevent unwanted cerebral ischemia in intensive care patients;Before each procedure applied to the patient, the amount of oxygen in the bloodstream circulating in the brain tissue should be constantly monitored. In the last guide published by the Brain Trauma Association;It is recommended that partial carbon dioxide pressure(PaCO2) is 35-40 mmHg, partial oxygen pressure(PaO2) is above 60 mmHg, and arterial oxygen saturation is 90% and above.In order to preserve these values, the patients are followed up in the mechanical ventilator for a while in the first period they exit the operation.

While the fact that the patients are connected to the mechanical ventilator may provide advantage in terms of providing continuous oxygenation,it may bring additional risks for the patients. Because the endotracheal suctioning suctioning need arises in the patient in the mechanical ventilator.There are important risks of endotracheal suctioning of mechanically ventilated patients with artificial in patients receiving mechanical ventilator support to prevent hypercarbia and hypoxia caused by secretion accumulated in the respiratory tract.These risks include hypoxia, arrhythmia, increase in MPD,hypertension,hypotension,agitation,pain,etc. countable.Especially during endotracheal suctioning, the increase of intracranial pressure in the patient, then the cough reflex induced and the high course of intracranial pressure after suctioning will disrupt cerebral perfusion,thus oxygenation of the brain is endangered.While blood flow and perfusion may be normal before and during the procedure,it changes to critical value afterwards and if it lasts more than 30 minutes,it poses a threat to patients.The position of the patient and the length of stay in the same position affect the cerebral circulation,reducing SPB.In this case,if the nursing follow-ups are insufficient or the attempts to protect the SME are ineffective;it becomes difficult for the brain to perform its functions, and even becomes unable to perform.

In the intensive care units,raising the head and positioning is a routine nursing initiative in order to protect patients from KIB and cerebral complications that may occur due to KIB.Different head heights and body positions applied after the neurosurgical intervention have been observed to affect secondary complications by affecting SME, PB and SKA.According to researches; lateral position given by raising the head of the bed, long-term flexion and extension of the head, the head being constantly 45° high are positions that may be harmful for neurosurgical patients.In addition, it has been reported that rotating or repositioning causes more secondary brain damage(7%) by increasing the ICU compared to other nursing interventions applied to patients. Secondary brain damage may result from 5 minutes after nursing interventions or more than 10 minutes from the beginning of nursing intervention,20 mmHg above KIB,60 mmHg below SPB,and 100 mmHg below systolic blood pressure. Responsibility of neurosurgical nurses;It is the safest way to provide the care that the patient needs without experiencing any undesirable side effects and secondary complications (respiratory events,cerebral ischemia,increased ICP,arrhythmia, etc.).This is directly related to the quality of the treatments. The results of the research showed that nurses should follow the cerebral oxygenation with non-invasive technique by constantly moving away from the invasive methods that cause many complications such as infection,arrhythmia,vascular injury to patients in the neurosurgery intensive care unit.

Since the oxygenation status of intensive care patients is measured and monitored with a pulse oximeter,the hypoxia state occurring in oxygenation in the brain tissue cannot be detected early. Standard methods used in the measurement of cerebral oxygenation have significant limitations in these patients.Jugular venous bulb oximetry measurement is an expensive method that requires invasive procedure;there is a risk of many complications such as infection on the patient, risk of tissue integrity deterioration,vascular injuries during bleeding of the catheter,bleeding; assessment of the measurement is essential by neurosurgeons;In addition, this method may miss regional ischemia.Non-invasive techniques such as transcranial doppler ultrasonography or electroencephalography(EEG) are other methods used indirectly to assess the adequacy of cerebral blood flow or the presence of ischemia.However,transcranial doppler and EEG are difficult to interpret by non-specialists. Cerebral oximetry device that measures oxygenation of the brain;It is important because it is a non-invasive method that monitors changes in cerebral oxygen metabolism,can provide continuous at the bedside, provides accurate and precise results as well as invasive methods,can provide nurses the convenience of interpretation independently in order not to cause secondary complications in nursing applications.Therefore,it can be easily evaluated in terms of nurses who are able to provide reliable and real-time data from several areas of the brain simultaneously, which is effective for the prevention and early detection of secondary injuries such as re-bleeding, vasospasm,cerebral ischemia,cerebral edema and seizure,and for 24 hours of patients.Cerebral oximetry device that works with near infrared spectroscopy(NIRS) technology,which can be used as a bedside monitor, is considered to be the most suitable device for patients and healthcare workers.

Studies have argued that low values in cerebral oximetry follow-ups may be predictors of hypoxic ischemic damage.In feasibility studies for the use of NIRS technology of neurocognitive and neurological complications during and after cardiac surgery;According to the transcranial doppler device of the cerebral oximeter device in adult patients;The use of this device has been suggested due to its advantages such as easy and uncomplicated use,clear,undoubtedly identifiable brain oxygenation, and nurses can evaluate independently.In studies, low regional regional oxygen level(rSO2) was directly and significantly interpreted with poor results after brain injury. In one study, the measurement of cerebral oxygen and hemoglobin values after vasospasm after subarachnoid hemorrhage was done with transcranial doppler and NIRS and its correlation with cortical ischemia was examined. Transcranial doppler failed to detect vasospasm in four of the six cases, while NIRS detected changes in the brain cortex and basal vessels.In the study,it was reported that a decrease of 3.9-6.4% compared to the basal value occurring in regional oxygenation was cut-off values predicting high sensitivity(100%) and specificity(85.7%) vasospasm.

When the literature is examined; Evidence that cerebral oxygenation monitoring is important in preventing complications such as delayed cerebral ischemia is clear. However, there is no evidence of the head height to be given during endotracheal suctioning and how long the head should remain in this position by affecting cerebral blood flow and KIB,which plays an important role in oxygenation of the brain.In a study,it is desired that the head height of neurosurgery patients should be 30 ° in terms of cerebral perfusion and should not exceed the 45 degree angle. Ledwith et al. (2010) also reported that the head height of 30 degrees in the supine position decreases CRB. Coşkun et al. (2011), in patients with cerebral vascular disease who did not undergo surgical intervention, they observed tracheal suctioning with a head height of only 15 and 30 degrees, and an increase in cerebral blood flow with a head height of 15 degrees in the measurement performed with transcranial doppler 5 minutes after the applicationWhen the intracranial pressure is continuously high for more than 30 minutes, SPB will deteriorate and the cerebral flow will be interrupted.In randomized controlled studies,it has been reported that adequate cerebral perfusion is provided at head heights up to 15 degrees and 60 degrees, but the ideal head height specified as 15° and 60° is very it remained uncertain in a wide range. In the results of the meta-analysis study, it was reported that the most suitable head height in terms of serabral perfusion was 30 and 45 degrees from 0,15,30 and 45 degrees in patients who underwent neurosurgery. However,it has been emphasized that the results related to the ideal head height are still contradictory in situations related to position change and other applications. In one study, when the head height was reduced from 30 degrees to 0 degrees in patients with head injuries, when the cerebral perfusion change was measured with NIRS technology; Cerebral perfusion pressure showed a significant change during the reduction of head height (p <0.001) and it was observed that the level of cerebral perfusion and oxy-hemoglobin increased by decreasing the head height. Although medical and nursing studies on this subject are still continuing today, there is no study investigating the effect of the ideal head height that should be within 30 minutes required for stabilization of cerebral perfusion and oxygenation during and after endotracheal suctioning.

There are no studies on the use of NIRS technology in nursing applications for neurosurgical patients. Brogan et al. (2017) 's systematic review and metaanalysis study; It was emphasized that studies examining the benefits of this technology in patients with traumatic brain injury are insufficient, and that both doctors and nurses should prove the benefits of this technology before and inside the hospital by conducting experimental research. In a study in which cost analysis was performed in patients who were followed up using NIRS technology;It was determined that there was an average decrease of 1937 dollars per patient (p=0.036) and it was pointed out that NIRS is a sensitive and reliable monitoring tool that eliminates the need for special nursing care. In line with these results,it is predicted that the nurses who are with the patient for 24 hours and who participate in the care and treatment of the patient can provide significant benefits for the patient by using this technology.With the simple use of this technology by nurses in intensive care settings, it is aimed to prevent many problems that may occur in patients and it is also thought that it will be cost-effective in patients with long hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Having undergone neurosurgery surgery,
* To get mechanical ventilator support,
* To have completed at least 6 hours in the mechanical ventilator, but not yet in the 72 hours,
* Being at the age of 18 and over,
* Life signs are stable (arterial blood pressure 160/90 mmHg; heart rate 70-100 / min, respiratory rate 16-20 / min, body temperature 36-37.5 ° c) and no pulmonary problems, Oxygen saturation level measured by pulse oximeter to be 85% and above,
* Glaskow Coma Score (GKS) not being below 9E,
* Na +, K +, Cl-, Hb, Hct values are within the normal reference range,
* Not having contraindications for head and body positioning,
* Volunteering to participate in the research.

Exclusion Criteria:

* Having another surgery apart from neurosurgery surgery,
* Not getting mechanical ventilator support,
* The time spent in the mechanical ventilator is less than 6 hours and more than 72 hours,
* Being under the age of 18,
* Life signs are unstable and have a pulmonary problem,
* Oxygen saturation level measured by pulse oximetry below 85%
* To be under Glaskow Coma Score (GKS) 9E,
* Na +, K +, Cl-, Hb, Hct values should not be within the normal reference range,
* Being a contraindication case for head and body positioning,
* Not to volunteer to participate in the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Turkey linked to the Health Ministry in the Western Black Sea Region Zonguldak Ataturk State Hospital intensive care unit treatment and care made postoperative mechanical ventilation due to brain surgery all the patient population of the study (according to information from the hospital's information-processing unit 01.01.2018- An average of 520 patients underwent brain surgery between 31.12.2018). The sample of the research, according to the research results obtained from the literature; α = 0.05, 0.25 effect size was determined as 46 patients with 90% power. The research was designed to make repeated measurements in a single group. Patients who meet the inclusion criteria will be included in the study.
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
To monitor the change of endotracheal suctioning in cerebral oxygenation parameter with non-invasive monitor in neurosurgery intensive care patients and to look at the statistical significance of the change. | The measurement will start with recording the value before the endotracheal suctıonıng application and end with recording the value at 30 minutes after the application. Results will be determined after reporting at the end of 1 year.
  Preservation of neurosurgical patients' cerebral perfusion is very important for the prognosis of patients. It is known that endotracheal aspiration,which is one of the nursing care practices applied in the intensive care follow-up of these patients,impairs the cerebral perfusions.However, although it is known, it is not sufficient to monitor the parameters showing the srebral perfusion status by the nurses who are constantly present with the patient.This parameter will be monitored with the regional oximeter device,which is considered to be the most accurate and appropriate method during and after endotracheal aspiration,which is one of the applications that change the cerebral perfusion status the most.In the literature, follow-up up to 30 minutes was planned, as the time required to correct cerebral perfusion was reported as 30 minutes in these patients

SECONDARY OUTCOMES:
To look at the effect of using technology for early diagnosis of complications such as cerebral ischemia in neurosurgery intensive care patients. | 1 year
  Changes in cerebral oxygenation may be an early sign of delayed complication of cerebral ischemia. Therefore, it is important to monitor the change in cerebral oxygenation. However, it is important that the best approach for monitoring this parameter is that patients can be monitored and evaluated by non-invasive healthcare professionals nurses, who are uninterrupted with the patients without leaving the intensive care environment. Therefore, the widespread use of such devices, which have proven their validity and reliability by using technology, suggests that the prognosis of the patients will have a good effect. Clinical research is needed for this. For this reason, in this group, which is a risky group, it is necessary to benefit from the technologies that non-invasive methods can be used without moving patients from their beds.
To determine the effect of endotracheal aspiration on 15% head height in cerebral oxygenation in neurosurgery intensive care patients. | 1 year
  Endotracheal aspiration application applied to patients disrupts the cerebral perfusion of patients. However, the impaired cerebral perfusion is expected to stabilize after application. If the time it takes for perfusion to return to normal exceeds 30 minutes, neuron damage begins to occur. During this period, the percentage of cerebral oxygenation, which is the parameter that shows the status of cerebral perfusion, should be monitored and necessary nursing care procedures should be carried out in order to stabilize. One application is to keep the head height of the patients at an appropriate angle. The ideal head height for this subject, which is a controversial subject in the literature and which is not yet talked about as evidence, is unknown. Clinical research is needed to examine the effect of 15 degrees of head height. Therefore, this is one of the results of this research.
To determine the effect of endotracheal aspiration procedure applied at 30 degree head height on the percentage of cerebral oxygenation in neurosurgery intensive care patients. | 1 year
  Endotracheal aspiration application applied to patients disrupts the cerebral perfusion of patients. However, the impaired cerebral perfusion is expected to stabilize after application. If the time it takes for perfusion to return to normal exceeds 30 minutes, neuron damage begins to occur. During this period, the percentage of cerebral oxygenation, which is the parameter that shows the status of cerebral perfusion, should be monitored and necessary nursing care procedures should be carried out in order to stabilize. One application is to keep the head height of the patients at an appropriate angle. The ideal head height for this subject, which is a controversial subject in the literature and which is not yet talked about as evidence, is unknown. Clinical research is needed to examine the effect of 30 degrees of head height. Therefore, this is one of the results of this research.
To determine the effect of endotracheal aspiration on 45% head height in cerebral oxygenation in neurosurgery intensive care patients. | 1 year
  Endotracheal aspiration application applied to patients disrupts the cerebral perfusion of patients. However, the impaired cerebral perfusion is expected to stabilize after application. If the time it takes for perfusion to return to normal exceeds 30 minutes, neuron damage begins to occur. During this period, the percentage of cerebral oxygenation, which is the parameter that shows the status of cerebral perfusion, should be monitored and necessary nursing care procedures should be carried out in order to stabilize. One application is to keep the head height of the patients at an appropriate angle. The ideal head height for this subject, which is a controversial subject in the literature and which is not yet talked about as evidence, is unknown. Clinical research is needed to examine the effect of 45 degrees of head height. Therefore, this is one of the results of this research.
The effect of age,gender,diagnosis, number of hospitalization days,mechanical ventilatory mode, glaskow coma scale score variables on patients' cerebral oxygenation before and after endotracheal suctionıng in patients with mechanical ventilation | 1 year
  Personal characteristics of the harvests related to the sociodemographic health status affect the general condition of the patients. The effect of endotracheal aspiration procedure applied to patients on cerebral oxygenation varies depending on these variables. Examining the direction of this effect is among the results of the research.

CONTACTS AND LOCATIONS:
Overall Officials: Zonguldak Bülent Ecevit University Faculty of Health Sciences, Principal Investigator — Zonguldak Bülent Ecevit University Faculty of Health Sciences
Locations (2):
- Turkey (Türkiye) (2):
  - Zonguldak Bülent Ecevit University Health Practice and Research Hospital, Zonguldak, Kozlu
  - Zonguldak Atatürk State Hospital, Zonguldak, Meşrutiyet

IPD SHARING:
Plan to Share IPD: Yes
All data ready to be published as a result of the research will be shared.
Time Frame: It will be available once the research is complete and ready for publication. There is no limit for the date of access.
Access Criteria: Completion and reporting of the study